CLINICAL TRIAL: NCT04972422
Title: A Phase 1b Study of ZN-c3 as a Single Agent in Patients With Solid Tumors
Brief Title: A Phase 1b Study of ZN-c3 in Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zentera Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: c3ZTCN100
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumors
Keywords: Solid Tumors
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Agent Dose Escalation (Experimental): Participants with solid tumors with advanced or metastatic disease who are refractory or ineligible to standard therapy(ies) or for whom no standard therapy is available.
  Interventions: Drug: ZN-c3

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 is a study drug
  Other Names: Study Drug

SUMMARY:
This is a Phase 1b open-label, multicenter study, evaluating the safety, tolerability, efficacy, pharmacokinetics (PK) and pharmacodynamics of ZN c3.

DETAILED DESCRIPTION:
This study consists of Dose Escalation and Dose Expansion component in Chinese subjects with solid tumors, described briefly as follows:

Dose Escalation: Single Agent Dose Escalation of ZN-c3 in solid tumors.

Dose Expansion: Single Agent ZN-c3 in solid tumors at the RP2D dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to initiation of any study-related procedures that are not considered standard of care.
2. Age ≥ 18 years or the minimum legal adult age (whichever is greater) at the time of informed consent.
3. Adequate hematologic and organ function as defined by the following criteria:

   1. ANC ≥ 1.5 × 109/L; excluding measurements obtained within 7 days after daily administration of filgrastim/sargramostim or within 3 weeks after administration of pegfilgrastim.
   2. Platelet count ≥ 100 × 109/L; excluding measurements obtained within 3 days after transfusion of platelets.
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastases, AST and ALT ≤ 5 x ULN.
   4. Total serum bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN in the case of Gilbert's disease.
   5. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 mL/min.
4. Female subjects of childbearing potential must have a negative serum beta human chorionic gonadotropin test.
5. Male subjects and female subjects of childbearing potential must agree to use an effective method of contraception per institutional standard prior to the first dose and for 90 days after the last dose of ZN-c3.
6. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
7. Willingness to practice adequate sun protection (use of sunscreen or sun-protective clothing or limitation of sun exposure).
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. Subjects must have a solid tumor with advanced or metastatic disease, refractory to standard therapy or for whom no standard therapy is available, or the subject is ineligible for standard therapy(ies).
10. Measurable or evaluable disease per RECIST version 1.1.
11. Subjects with advanced or metastatic disease, refractory to standard therapy or for whom no standard therapy is available, or the subject is ineligible for standard therapy(ies).

Exclusion Criteria:

1. Any of the following treatment interventions within the specified time frame prior to Cycle 1 Day 1:

   1. Major surgery within 28 days (the surgical incision should be fully healed prior to study drug administration).
   2. Radiation therapy within 21 days; however, if the radiation portal covered ≤ 5% of the bone marrow reserve, the subject is eligible irrespective of the end date of radiotherapy.
   3. Any prior systemic therapy regardless of the stop date, but the subject must have recovered to eligibility levels from prior toxicity.
   4. Autologous or allogeneic stem cell transplant within 3 months.
   5. Current use of an investigational agent that is not expected to be cleared by the first dosing of study drug or that has demonstrated to have prolonged side effects. Subjects should have recovered from the side effects to a Grade 0 or 1 (except alopecia).
2. A serious illness or medical condition(s) including, but not limited to, the following:

   1. Brain metastases that require immediate treatment or are clinically or radiologically unstable (i.e., have been stable for < 1 month). If receiving steroids, subjects must be receiving a stable to decreasing corticosteroid dose during at least 1 week before enrollment.
   2. Leptomeningeal disease that requires or is anticipated to require immediate treatment.
   3. Myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV).
   4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the subject inappropriate for entry into this study.
   5. Significant gastrointestinal abnormalities, including an inability to take oral medication, requirement for IV alimentation, active peptic ulcer, chronic diarrhea or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption.
   6. Active or uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥ 72 hours.
3. Unresolved toxicity of Grade > 1 attributed to any prior therapies (excluding Grade 2 neuropathy, alopecia or skin pigmentation).
4. Prior therapy with ZN-c3 or known hypersensitivity to any drugs similar to ZN c3 in class.
5. Prior therapy with a WEE1 inhibitor.
6. Pregnant or lactating females (including the cessation of lactation) or females of childbearing potential who have a positive serum pregnancy test within 14 days prior to Cycle 1 Day 1.
7. Subjects with active (uncontrolled, metastatic) second malignancies or requiring therapy.
8. Individuals who are judged by the Investigator to be unsuitable as study subjects.
9. 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of > 450 msec, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.
10. History or current evidence of congenital long QT syndrome.
11. Administration of strong and moderate CYP3A4 inhibitors and inducers as well as strong and moderate P-gp inhibitors.
12. Patients with active HBV and HCV infection: HBV DNA is higher than the upper limit of reference value if anti-HBC positive, HCV virus copy number exceeds the lower limit of detection method.
13. A known history of human immunodeficiency virus infection or serum anti-HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Until 30 days after the last dose of study drug
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Incidence and severity of dose-limiting toxicities (DLTs) in DLT evaluable subjects during Cycle 1 | At the end of Cycle 1 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Sichuan University Huaxi Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided